CLINICAL TRIAL: NCT03772119
Title: Assessment and Follow-up of Surgical Treatment of Hemivertebra in Children
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI17/HEMIVERTEBRE SOFOP
Record Dates: First submitted 2018-11-22; First posted 2018-12-11 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Hemivertebra
Keywords: Vertebral Malformation; Hemivertebra; Surgical resection; SOFOP

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical treatment of hemivertebra: cohort of children with a vertebral malformation treated by surgical resection
  Interventions: Procedure: Surgical resection

INTERVENTIONS:
Procedure: Surgical resection — Surgical resection of hemivertebra

SUMMARY:
The treatment of child's vertebral malformations has evolved a lot including the realization of surgical vertebral resections. The surgical techniques used are multiple, require heavy surgery, one or more approaches and surgical time, transfusions, a neurological risk (up to 20% in some series, risk of non-consolidation, insufficient correction). These surgical techniques deserve an evaluation of the early complications and the skeletal maturity of these children (maintenance of the surgical correction, evolution of the associated curvatures).

DETAILED DESCRIPTION:
The treatment of child's vertebral malformations has evolved a lot including the realization of surgical vertebral resections. The surgical techniques used are multiple, require heavy surgery, one or more approaches and surgical time, transfusions, a neurological risk (up to 20% in some series, risk of non-consolidation, insufficient correction). These surgical techniques deserve an evaluation of the early complications and the skeletal maturity of these children (maintenance of the surgical correction, evolution of the associated curvatures).

ELIGIBILITY:
Inclusion Criteria:

* Child from 3 to 10 years old
* with a vertebral malformation requiring surgery for hemivertebras

Exclusion Criteria:

* Child previously operated on the spine
* Different procedure of a surgical resection of vertebral malformation
* Absence of medical follow-up
* Parents refusal concerning data storage

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children from 3 to 10 years old with vertebral malformation requiring surgery for hemivertebra
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-02-04 (Actual); Primary Completion 2039-02 (Estimated); Study Completion 2039-02 (Estimated)

PRIMARY OUTCOMES:
Immediate effectiveness of surgery: Evolution of Cobb angle | From baseline to 6 months after surgery
  Effectiveness of immediate correction : spinal deformities measured by the Cobb angle on radios face and profile
Appearances of complications | From baseline to 6 months after surgery
  Appearances of complications (neurological, vascular, non consolidation) at 6 months. These complications will be gathered from hospitalization reports.
Late persistence of complications | From 6 months after surgery to 15 years
  Persistent complications will be collected through clinical examination at follow-up visits.

SECONDARY OUTCOMES:
Long-term effectiveness of surgery: Evolution of Cobb angle | From 6 months after surgery to 15 years
  Maintaining local correction with growth: spinal deformities measured by the Cobb angle on radios face and profile

CONTACTS AND LOCATIONS:
Overall Officials: Thierry ODENT, MD-PhD, Study Director — University Hospttal, Tours
Locations (13):
- France (13):
  - Pediatric Surgery Service, University Hospital, Bordeaux, Bordeaux
  - Pediatric Surgery Service, University Hospital, Grenoble, Grenoble
  - Pediatric Surgery Service, University Hospital, Lyon, Lyon
  - Pediatric Surgery Service, University Hospital, Marseille, Marseille
  - Pediatric Surgery Service, University Hospital, Nantes, Nantes
  - Pediatric Surgery Service, University Hospital, Nice, Nice
  - Pediatric Surgery Service, University Hospital, Armand Trousseau Hospital, AP-HP, Paris
  - Pediatric Surgery Service, Robert-Debré Hospital, AP-HP, Paris
  - Pediatric Surgery Service, University Hospital, Necker Hospital, AP-HP, Paris
  - Pediatric Surgery Service, University Hospital, Rennes, Rennes
  - Pediatric Surgery Service, University Hospital, Saint-Etienne, Saint-Etienne
  - Pediatric Surgery Service, University Hospital, Toulouse, Toulouse
  - Pediatric Surgery Service, University Hospital, Tours, Tours

IPD SHARING:
Plan to Share IPD: No